CLINICAL TRIAL: NCT02183558
Title: Glucose Metabolism and Screening for Gestational Diabetes Mellitus According to Different Sets of Criteria in Women With Polycystic Ovary Syndrome and Controls
Brief Title: Screening for GDM in Women With PCOS and Controls
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Region of Southern Denmark (Other); Municipality of Odense (Other Government); University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Marianne Andersen, DMSci, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: GDM OBK; Glucose OBK (Other: Odense University Hospital)
Record Dates: First submitted 2014-06-20; First posted 2014-07-08 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Polycystic Ovary Syndrome; Gestational Diabetes Mellitus
Keywords: PCOS; GDM; OGTT; Glucose metabolism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- OGTT by randomization (Experimental): Women without risk factors for GDM are offered OGTT in gestational week 28
  Interventions: Other: OGTT by randomization
- OGTT by indication (Experimental): Women with risk factors for OGTT are offered diagnostic 2 hour OGTT in pregnancy week 28
  Interventions: Other: OGTT by indication

INTERVENTIONS:
Other: OGTT by randomization
  Arms: OGTT by randomization
Other: OGTT by indication
  Arms: OGTT by indication

SUMMARY:
Women with polycystic ovary syndrome (PCOS) are often insulin resistant. During pregnancy, insulin sensitivity decreases. The investigators examine glucose metabolism during oral glucose tolerance test and the incidense of gestational diabetes mellitus in a prospective cohort of pregnant women with PCOS and controls.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy achieved during 2010-2012
* Residents of the municipality of Odense

Exclusion Criteria:

* Moving from Odense during pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2500 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Gestational diabetes mellitus | 2 years
  Gestational diabetes mellitus diagnosed by oral glucose tolerance test in gestational week 28 in women with and without risk factors for gestational diabetes mellitus.
Gestational Diabetes Mellitus | Gestational week 28
  Gestational diabetes mellitus is diagnosed by 2 hour 75 gram oral glucose tolerance test in gestational week 28

SECONDARY OUTCOMES:
Anthropometric measures in offspring | At birth
  The association between blood glucose values and anthropometric measures (birth length, weight and abdominal circumference) at birth in the offspring is investigated

CONTACTS AND LOCATIONS:
Overall Officials: Marianne Andersen, DMSci, Principal Investigator — Odense University Hospital
Locations (1):
- OdenseUH, Odense, Denmark

REFERENCES:
- [Derived] Al-Jorani H, Jensen RC, Jensen TK, Christesen HT, Jorgensen JS, Bacmeister L, Dechend R, Glintborg D, Jensen BL, Andersen MS. Diurnal Urinary Aldosterone Excretion and Potassium Intake During Pregnancy Are Associated With High Normal Blood Pressure in Early Childhood. J Am Heart Assoc. 2025 Jul 15;14(14):eJAHA2025042165T. doi: 10.1161/JAHA.124.042165. Epub 2025 Jul 3. PMID 40611483